CLINICAL TRIAL: NCT05373277
Title: KF2019#1-tutkimus: Verihiutaleiden estäjän Vaikutus kolesterolilääkkeeseen
Brief Title: KF2019#1-trial: Effects of a Thrombocyte Inhibitor on a Cholesterol-lowering Drug
Acronym: KF2019#1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Mikko Niemi, Professor, head physician, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KF2019#1
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ticagrelor; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The subjects will be given orally placebo twice a day for 2 days, and a single 10 mg dose of rosuvastatin.
  Interventions: Drug: Placebo; Drug: Rosuvastatin
- Ticagrelor (Active Comparator): The subjects will be given orally 90 mg ticagrelor twice a day for 2 days, and a single 10 mg dose of rosuvastatin.
  Interventions: Drug: Ticagrelor; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Placebo — one tablet of placebo twice daily for two days
  Arms: Placebo
Drug: Ticagrelor — Intervention Description: 90 mg tablet twice daily for two days
  Arms: Ticagrelor
Drug: Rosuvastatin — 10 mg tablet, single dose

SUMMARY:
The cholesterol-lowering drug rosuvastatin is a substrate of the breast cancer resistance protein (BCRP). BCRP is an efflux transporter expressed e.g. in the small intestine. It limits the oral bioavailability of rosuvastatin by transporting rosuvastatin from enterocytes back to the gut lumen. Inhibition of BCRP can increase rosuvastatin bioavailability and systemic concentrations. Ticagrelor is a platelet aggregation inhibitor used in treatment and prevention of atherothrombotic events. Ticagrelor may inhibit BCRP in humans. This study is aimed to investigate the possible interaction of rosuvastatin with ticagrelor. Ten healthy male or female non-smoking volunteers aged 18-40 years are taken into the study. Primary endpoint is area under the plasma concentration-time curve of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-40
* Healthy
* Systolic blood pressure ≥100 mmHg
* Accepted results from laboratory tests (blood haemoglobin, basic blood count and blood platelets, alanine aminotransferase, alkaline phosphatase, glutamyl transferase, creatinine, plasma potassium and sodium). Negative pregnancy test result (serum human chorionic gonadotropin) for women.
* Fully vaccinated against COVID-19.

Exclusion Criteria:

* Significant disease
* Abnormal result from the Helsinki University Hospital bleeding questionnaire
* Smoking
* Using oral contraception pills or other regular medication
* Pregnancy (current or planned) or nursing
* Participation in any other studies involving investigational or marketed drug products within three months prior to the entry into this study
* Donation of blood within three months prior to the entry into this study
* Significant overweight / small or hard-to-find veins
* Weight < 45 kg
* BMI < 18.5 kg/m2
* Insufficient Finnish language skills

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-11 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration - time curve of rosuvastatin | Prior to and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 23, and 47 hours after administration of rosuvastatin

SECONDARY OUTCOMES:
Peak plasma concentration, half-life, time to peak plasma concentration, amount excreted, and renal clearance of rosuvastatin | Prior to and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 23, and 47 hours after administration of rosuvastatin

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No